CLINICAL TRIAL: NCT03352674
Title: Open Label Randomized Multicenter Clinical Trial to Compare Immunogenicity of Insulin Glargine Ezelin vs Lantus in Type 2 Diabetes Mellitus Patients
Brief Title: Immunogenicity Study of Insulin Glargine Ezelin vs Lantus in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr Tri Juli Edi Tarigan, SpPD-KEMD, Endocrinologist, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaU-01
Record Dates: First submitted 2017-10-14; First posted 2017-11-24 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus
Keywords: insulin glargine; diabetes mellitus; immunogenicity
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin Glargine Ezelin (Experimental): Drug product Insulin Glargine, Ezelin 100 U/mL (PT Kalbe Farma, Tbk)
  Interventions: Drug: Insulin Glargine Ezelin
- Insulin Glargine Lantus (Active Comparator): Insulin Glargine Pen Injector [Lantus]
  Interventions: Drug: Insulin Glargine Pen Injector [Lantus]

INTERVENTIONS:
Drug: Insulin Glargine Ezelin — Insulin Glargine (Ezelin) once daily at individually adjusted dose
  Other Names: Ezelin
  Arms: Insulin Glargine Ezelin
Drug: Insulin Glargine Pen Injector [Lantus] — Insulin Glargine (Lantus) once daily at individually adjusted dose
  Other Names: Lantus
  Arms: Insulin Glargine Lantus

SUMMARY:
This is an open-label randomised multicenter clinical study to compare immunogenicity of the drug products Insulin Glargine (Kalbe Farma) and Lantus (Sanofi -Aventis) in type 2 diabetes mellitus patients

DETAILED DESCRIPTION:
Previous study has revealed that Insulin Glargine (Kalbe Farma) has similar efficacy with Lantus (Sanofi-Aventis) in controlling blood glucose in type 2 diabetes mellitus patients, but the immunogenicity potential of this product has not been known. Therefore, the present study is aiming to compare immunogenicity of Insulin Glargine (Kalbe Farma) and Lantus (Sanofi-Aventis) in type 2 diabetes mellitus patients in an open-label randomised multicenter clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18 years old and above
* Diabetes mellitus type 2 patients who has failed an oral hypoglycemic drug products, insulin-naive, disease duration of at least 6 months, inadequate glycemic control (HbA1c > 7.0 %)
* BMI ranged from 19 - 35 kg/m2
* Consent from patients of childbearing potential to use contraception method throughout the study
* Signed informed consent form

Exclusion Criteria:

* History of diabetic ketoacidosis more than 2 times in the past 1 year
* History of pancreatectomy
* Estimated glomerular filtration rate <30 mL/min
* Positive ZnT8 Antibody
* Treatment with glucocorticoids, immunodepressant or cytostatics in 60 days before study.
* Any malignant disease, including in medical history
* Drugs and alcohol abuse, including in medical history
* Hipersensitivity to insulin glargine or any excipient of the drugs from medical history
* Mental disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of immune response | 6 months
  Production of antibodies against insulin /IAA and ZnT8 antibody in investigational drug product and comparator groups

SECONDARY OUTCOMES:
HbA1c | 6 months
  change in HbA1c level after 6 months of therapy compared to baseline value
Fasting blood glucose | 6 months
  Change in fasting blood glucose
Hypoglycemia | 6 months
  Incidence and severity of hypoglycaemia cases
Adverse events | 6 months
  Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tri Juli Edi Tarigan, MD, Principal Investigator — Cipto Mangunkusumo Hospital/Faculty of Medicine Universities Indonesia
Locations (1):
- Department of Internal Medicine Cipto Mangunkusumo Hospital, Faculty of Medicine Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chakkarwar PN, Manjrekar NA. Insulin glargine: a long acting insulin analog. J Postgrad Med. 2005 Jan-Mar;51(1):68-71. PMID 15793346
- [Result] McKeage K, Goa KL. Insulin glargine: a review of its therapeutic use as a long-acting agent for the management of type 1 and 2 diabetes mellitus. Drugs. 2001;61(11):1599-624. doi: 10.2165/00003495-200161110-00007. PMID 11577797
- [Result] Garber AJ, Abrahamson MJ, Barzilay JI, Blonde L, Bloomgarden ZT, Bush MA, Dagogo-Jack S, Davidson MB, Einhorn D, Garvey WT, Grunberger G, Handelsman Y, Hirsch IB, Jellinger PS, McGill JB, Mechanick JI, Rosenblit PD, Umpierrez G, Davidson MH; American Association of Clinical Endocrinologists. AACE comprehensive diabetes management algorithm 2013. Endocr Pract. 2013 Mar-Apr;19(2):327-36. doi: 10.4158/endp.19.2.a38267720403k242. No abstract available. PMID 23598536
- [Result] Pihoker C, Gilliam LK, Hampe CS, Lernmark A. Autoantibodies in diabetes. Diabetes. 2005 Dec;54 Suppl 2:S52-61. doi: 10.2337/diabetes.54.suppl_2.s52. PMID 16306341
- [Result] Bingley PJ. Clinical applications of diabetes antibody testing. J Clin Endocrinol Metab. 2010 Jan;95(1):25-33. doi: 10.1210/jc.2009-1365. Epub 2009 Oct 29. PMID 19875480
- [Result] Vaziri-Sani F, Oak S, Radtke J, Lernmark K, Lynch K, Agardh CD, Cilio CM, Lethagen AL, Ortqvist E, Landin-Olsson M, Torn C, Hampe CS. ZnT8 autoantibody titers in type 1 diabetes patients decline rapidly after clinical onset. Autoimmunity. 2010 Dec;43(8):598-606. doi: 10.3109/08916930903555927. Epub 2010 Mar 19. PMID 20298127
- [Result] Pan CY, Sinnassamy P, Chung KD, Kim KW; LEAD Study Investigators Group. Insulin glargine versus NPH insulin therapy in Asian Type 2 diabetes patients. Diabetes Res Clin Pract. 2007 Apr;76(1):111-8. doi: 10.1016/j.diabres.2006.08.012. Epub 2006 Oct 2. PMID 17011662
- [Result] Rosenstock J, Dailey G, Massi-Benedetti M, Fritsche A, Lin Z, Salzman A. Reduced hypoglycemia risk with insulin glargine: a meta-analysis comparing insulin glargine with human NPH insulin in type 2 diabetes. Diabetes Care. 2005 Apr;28(4):950-5. doi: 10.2337/diacare.28.4.950. PMID 15793205
- [Result] Rosenstock J, Davies M, Home PD, Larsen J, Koenen C, Schernthaner G. A randomised, 52-week, treat-to-target trial comparing insulin detemir with insulin glargine when administered as add-on to glucose-lowering drugs in insulin-naive people with type 2 diabetes. Diabetologia. 2008 Mar;51(3):408-16. doi: 10.1007/s00125-007-0911-x. Epub 2008 Jan 16. PMID 18204830
- [Result] Rosenstock J, Schwartz SL, Clark CM Jr, Park GD, Donley DW, Edwards MB. Basal insulin therapy in type 2 diabetes: 28-week comparison of insulin glargine (HOE 901) and NPH insulin. Diabetes Care. 2001 Apr;24(4):631-6. doi: 10.2337/diacare.24.4.631. PMID 11315821
- [Result] Stumvoll M, Goldstein BJ, van Haeften TW. Type 2 diabetes: principles of pathogenesis and therapy. Lancet. 2005 Apr 9-15;365(9467):1333-46. doi: 10.1016/S0140-6736(05)61032-X. PMID 15823385
- [Result] Rubin RR, Peyrot M, Siminerio LM. Health care and patient-reported outcomes: results of the cross-national Diabetes Attitudes, Wishes and Needs (DAWN) study. Diabetes Care. 2006 Jun;29(6):1249-55. doi: 10.2337/dc05-2494. PMID 16732004
- [Result] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Result] Yki-Jarvinen H, Juurinen L, Alvarsson M, Bystedt T, Caldwell I, Davies M, Lahdenpera S, Nijpels G, Vahatalo M. Initiate Insulin by Aggressive Titration and Education (INITIATE): a randomized study to compare initiation of insulin combination therapy in type 2 diabetic patients individually and in groups. Diabetes Care. 2007 Jun;30(6):1364-9. doi: 10.2337/dc06-1357. Epub 2007 Mar 23. PMID 17384341
- [Derived] Tarigan TJE, Dwijayanti A, Setyowati S, Louisa M. Immunogenicity and Efficacy of Insulin Glargine Biosimilar Ezelin versus Originator Insulin Glargine in Patients with Type 2 Diabetes. Diabetes Metab Syndr Obes. 2021 Jan 12;14:107-116. doi: 10.2147/DMSO.S279385. eCollection 2021. PMID 33469328